CLINICAL TRIAL: NCT01174017
Title: A Study Assessing the Ability of AnchorSeed Iodine-125 Sources to Hold Fast in Tissue When Implanted for Treatment of Localized Prostate Cancer
Brief Title: Ability of a New Design of Iodine 125 Seed to Maintain Intended Position When Implanted in the Prostate
Acronym: FAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Principal Investigator, Juanita Crook, MD, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-01685
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Iodine 125 brachytherapy; seed migration; seed migration in the first month after brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard loose Iodine 125 seeds (Active Comparator): Prostate brachytherapy implant to be performed with standard format loose Iodine 125 seeds
  Interventions: Radiation: Iodine 125 standard loose brachytherapy seeds
- AnchorSeed Iodine 125 implant (Experimental): Prostate brachytherapy implant to be performed with a new design of Iodine 125 seed that has a coating to increase adherence to tissue
  Interventions: Radiation: AnchorSeed Iodine 125 brachytherapy prostate implant

INTERVENTIONS:
Radiation: Iodine 125 standard loose brachytherapy seeds — radioactivity 0.4 U per seed, prescribed dose 144 Gy
  Other Names: BrachySciences
  Arms: Standard loose Iodine 125 seeds
Radiation: AnchorSeed Iodine 125 brachytherapy prostate implant — activity 0.4 U per seed, prescribed dose 144 Gy
  Other Names: BrachySciences
  Arms: AnchorSeed Iodine 125 implant

SUMMARY:
This study compares the ability of a new design of brachytherapy seed for prostate seed implants for treatment of prostate cancer to maintain their intended position in the prostate after being deposited. Standard seeds, especially in apical locations, have a tendency to migrate distally in response to muscular forces. AnchorSeeds have a textured coating which is designed to prevent migration. 40 patients who are eligible and suitable for prostate brachytherapy will be randomly assigned to receive either standard seeds or AnchorSeeds.

DETAILED DESCRIPTION:
Standard post implant prostate brachytherapy quality assurance at the Center for the Southern Interior is usually performed at one month after the procedure with CT and MR imaging. In order to test the ability of the new design of prostate brachytherapy seeds (AnchorSeeds) to hold their position in the prostate, 40 men who have been randomly assigned to receive either standard seeds or AnchorSeeds will have an additional CT scan immediately after the procedure to record seed position for comparison to positions one month later. The magnitude and frequency of seed displacement will be determined.

ELIGIBILITY:
Inclusion Criteria:

* localized prostate cancer
* favorable or intermediate risk
* suitable for permanent seed implant by functional and technical criteria

Exclusion Criteria:

* patient unwilling to have a second CT scan for study purposes
* claustrophobic patient unable to have CT scan
* patient unsuitable for brachytherapy because of prostate size or poor voiding function
* patient medically unable to stop anticoagulants for procedure

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
seed displacement | one month
  CT scan of the prostate immediately after the implant will be used to determine the center of mass of the implant as a reference for distal migration of apical seeds and compared to positions on the CT scan one month following the implant

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center for the Southern Interior, Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Badwan HO, Shanahan AE, Adams MA, Shanahan TG, Mueller PW, Markwell SJ, Tarter TH. AnchorSeed for the reduction of source movement in prostate brachytherapy with the Mick applicator implant technique. Brachytherapy. 2010 Jan-Mar;9(1):23-6. doi: 10.1016/j.brachy.2009.07.002. Epub 2009 Sep 17. PMID 19762286